CLINICAL TRIAL: NCT02456493
Title: The Effect of Carotid IMT (Intima Media Thickness) on Postoperative Cognitive Dysfunction in Patients Undergoing Off-Pump Coronary Artery Bypass Graft Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0254
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Occlusive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- increased carotid IMT group: Patients who have increased carotid IMT (intima media thickness)
- normal carotid IMT group: Patients who have normal carotid IMT

SUMMARY:
The patients who have undergone cardiac surgery have higher likelihood of postoperative cognitive dysfunction (POCD). The carotid intima-media thickness (IMT) is associated with cognitive dysfunction in the old. The aim of this study is to evaluate the effect of carotid IMT in patients undergoing OPCAB(off-pump coronary artery bypass surgery) on postoperative cognitive dysfunction. Two hundred twenty four patients, aged 20 to 79 years, scheduled for OPCAB will be divided into increased IMT (n=112) and normal IMT (n=112) group by preoperative B-mode ultrasonography. The cognitive function measured by K-MMSE, MOCA-K before the operation, and on the 7 day, 3 months after operation. The patients in the non-surgical group are measured three times: baseline, after 7days, after 3 months.

ELIGIBILITY:
Inclusion Criteria:

- patients who are scheduled to undergo OPCAB

Exclusion Criteria:

* severe cognitive dysfunction
* disabling mental change disorder
* unable to communicate or speak Korean
* do not have carotid IMT measurement.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are schedued to undergo OPCAB
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
postoperative cognitive dysfunction | 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea